CLINICAL TRIAL: NCT07169721
Title: CIRCAdian Rhythm of the IMMune Age IndeX (CIRCA-IMMAX) - Influence of Circadian Rhythm on the Determination of an Immune Age Metric
Brief Title: CIRCAdian Rhythm of the IMMune Age IndeX (IMMAX)
Acronym: CIRCA-IMMAX
Status: Completed | Type: Observational
Sponsor: Leibniz Research Centre for Working Environment and Human Factors (Other)
Responsible Party: Sponsor
Other Study IDs: Ethics committee approval: 243
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Healthy Subjects; Immune Cells (Mucosal and Systemic)
Keywords: immune age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the influence of circadian rhythms on the determination of an individual's immune age. The biomarker IMMAX was calculated for 50 participants aged 20-69 at 8 a.m., 1 p.m. and 6 p.m. on the same day.

ELIGIBILITY:
Inclusion Criteria:

* aged > 18 years
* knowledge of German or English sufficient to provide verbal explanations and obtain written consent

Exclusion Criteria:

* exercise on the assessment day
* acute infection
* vaccination within the last 4 weeks
* autoimmune disease
* cancer
* drugs that may influence immune cell counts
* participation in other interventional studies during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects who are willing to visit the study centre in Dortmund three times a day.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Changes in the Immune Age Index Immune Age Index (IMMAX) from morning to midday and evening | From 8 a.m. until 6 p.m. on the same day
  To determine the Immune Age Index, 100 µl blood is collected and immunostained with antibodies. The immune cells are then analyzed using flow cytometry. IMMAX values range from 0 to 1 with higher values indicating a higher immune age.

CONTACTS AND LOCATIONS:
Locations (1):
- Leibniz Research Centre for Working and Environment and Human Factors, Dortmund, Germany

REFERENCES:
- [Background] Brode P, Claus M, Gajewski PD, Getzmann S, Wascher E, Watzl C. From Immunosenescence to Aging Types-Establishing Reference Intervals for Immune Age Biomarkers by Centile Estimation. Int J Mol Sci. 2023 Aug 24;24(17):13186. doi: 10.3390/ijms241713186. PMID 37685992
- [Background] Brode P, Claus M, Gajewski PD, Getzmann S, Golka K, Hengstler JG, Wascher E, Watzl C. Calibrating a Comprehensive Immune Age Metric to Analyze the Cross Sectional Age-Related Decline in Cardiorespiratory Fitness. Biology (Basel). 2022 Oct 27;11(11):1576. doi: 10.3390/biology11111576. PMID 36358277